CLINICAL TRIAL: NCT01714804
Title: Efficacy and Safety of Integra Accell Evo3 Demineralized Bone Matrix in Instrumented Lumbar Spine Fusion
Brief Title: Efficacy and Safety of Integra Accell Evo3 DBM in Instrumented Lumbar Spine Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SeaSpine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACC3-US-2012-1
Record Dates: First submitted 2012-10-22; First posted 2012-10-26 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Stenosis; Spondylosis; Degenerative Changes
Keywords: Bone Morphogenetic Protein (BMP); Demineralized bone matrix (DBM); Fusion rates; Interbody fusion; Lumbar spine; Transverse lumbar interbody fusion (TLIF); Patient reported outcomes; Posterolateral lumbar fusion (PLF)
MeSH Terms: conditions — Constriction, Pathologic; Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prospective (Experimental): Accell Evo3
  Interventions: Device: Accell Evo3 Prospective Use

INTERVENTIONS:
Device: Accell Evo3 Prospective Use

SUMMARY:
The objective of this study is to prospectively evaluate the performance of Integra Accell Evo3 Demineralized Bone Matrix as an adjunct for instrumented lumbar spine fusion with a retrospective comparison to a historical patient cohort.

DETAILED DESCRIPTION:
The objective of this study is to prospectively evaluate the performance of Integra Accell Evo3 Demineralized Bone Matrix as an adjunct for instrumented lumbar spine fusion in comparison to a retrospective cohort of Infuse subjects. Infuse subjects were not enrolled in the current study.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 (eighteen) years of age or older at the time of surgery.
* Require spinal fusion using TLIF, PLF or PLIF, with the use of an interbody spacer, at 1 to 3 levels between L3-S1.
* Willing and able to return for the scheduled follow-up visits, follow post-operative instructions and undergo the required radiographic exams (A/P, Lateral Neutral and Lateral Flexion/Extension X-rays) for up to 3 time points between 6 months and 24 months post-surgery (6±2 months, 12±3 months and 24±4 months post-surgery), including one CT-scan at 12±3 months.
* Unresponsive to conservative care over a period of at least 6 months or has signs and/or symptoms that mandate urgent surgical intervention.

Exclusion Criteria:

* Are long term users of medications (i.e. steroids greater than 2-weeks) that are known to inhibit fusion or bone metabolism at any time within 6 months prior to surgery. Exceptions are inhaled steroids for asthma treatment (i.e. patients on inhaled steroids are allowed), or epidural steroid injections.
* Are taking immunosuppressive agents (Cancer chemotherapy, treatment with Disease Modifying Anti-rheumatic drugs (DMARDs) or any similar immunomodulating drugs) or are treated with Growth Factors or Insulin at any time within 6 months prior to surgery.
* Are being treated with radiotherapy.
* Are having medical conditions, known to impact bone metabolism, such as Paget's disease, osteoporosis.
* Are smokers and/or nicotine/tobacco users.
* Are pregnant, lactating or women wishing to become pregnant.
* Are a prisoner.
* Are currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the study endpoints.
* Prior spine surgery at the index level except posterior decompressive surgery where the posterior elements are preserved e.g. facet saving techniques such as discectomy, laminotomy, and intradiscal procedures.
* Use of any other bone graft or bone graft substitute in addition to or in place of Accell Evo3® with the exception of local autograft and/or cancellous bone chips.
* Use of routine prophylactic NSAIDS for 3 months post-operatively, but low dose concomitant pain medications e.g. aspirin should be continued and recorded on the Concomitant Pain Medications case report form (CRF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Youssef, MD, Principal Investigator — Spine Colorado
Locations (1):
- Spine Colorado, Durango, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Accell Evo3: Prospectively enrolled patients who required posterolateral fusion at one to three levels between L3 and S1. Treatment included standard instrumented posterolateral fusion with interbody fusion by TLIF at the discretion of the surgeon. Accell Evo3 was used with autogenous cancellous bone in the posterolateral space.
- Infuse: Retrospective patients who were treated with posterolateral fusion at one to three levels between L3 and S1. Treatment included standard instrumented posterolateral fusion with interbody fusion by TLIF at the discretion of the surgeon. Infuse (rh-BMP2) was used with autogenous cancellous bone in the posterolateral space. Subjects in this treatment arm were historical controls and were not enrolled in this study.
Period: Overall Study
Arm/Group | Accell Evo3 | Infuse
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prospective: Accell Evo3
  Accell Evo3 prospective study arm
- Retrospective: Infuse
  rh-BMP2 retrospective study arm
- Total: Total of all reporting groups
Arm/Group | Prospective | Retrospective | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Customized [Count of Participants; unit: Participants]
  >18 years old | 29 | 30 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 13 | 13 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Levels With Posterolateral Fusion
Description: Assessment of fusion in the posterolateral space was performed using by X-ray and/or CT. Assessment was performed by the operating surgeon blinded towards patient. Each spinal level was graded separately
Time Frame: 12 months
Population: One level is defined as a spinal segment in the lumbar spine.
Measure: Count of Units; unit: levels
Units Other Than Participants: levels
Groups:
- Accell Evo3: Prospectively enrolled patients who required posterolateral fusion at one to three levels between L3 to S1. Treatment included standard instrumented posterolateral fusion with interbody fusion by TLIF at the discretion of the surgeon. Accell Evo3 was used with autogenous cancellous bone in the posterolateral space.
- Infuse: Retrospective patients who were treated with posterolateral fusion at one to three levels between L3 to S1. Treatment included standard instrumented posterolateral fusion with interbody fusion by TLIF at the discretion of the surgeon. Infuse (rh-BMP2) was used with autogenous cancellous bone in the posterolateral space.
Arm/Group | Accell Evo3 | Infuse
Number analyzed (Participants) | 29 | 30
Number analyzed (levels) | 36 | 37
levels | 23 | 26

2. Secondary Outcome: Oswestry Disability Index (ODI), Visual Analog Scale (VAS) for Pain in the Back (VAS-back) and in the Leg (VAS-leg)
Time Frame: 12 months
Population: Data were not collected
Arm/Group | Accell Evo3 | Infuse
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months post surgery
Description: Adverse events: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research
Groups:
- Infuse: Retrospective patients who were treated with posterolateral fusion at one to three levels between L3 and S1. Treatment included standard instrumented posterolateral fusion with interbody fusion by TLIF at the discretion of the surgeon. Infuse (rh-BMP2) was used with autogenous cancellous bone in the posterolateral space.
Arm/Group | Accell Evo3 | Infuse
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 7/29 | 2/30
Other Adverse Events (participants affected / at risk) | 6/29 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Accell Evo3 (N=29) | Infuse (N=30)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
epidural hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Adjacent segment disease (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Blood Pressure increase (Cardiac disorders) | 1 (1) | 0 (0)
Cataract surgery (Eye disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
carpal tunnel trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CMC arthroplasty, thumb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
headache, rib and back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper extremity numbness; guyon's canal release (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Surgery for lipoma, right flank (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Accell Evo3 (N=29) | Infuse (N=30)
Back and thigh pain (stinging) (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Numbness (Nervous system disorders) | 2 (2) | 0 (0)
Fever and burning around incision (Infections and infestations) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Adjacent segment disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria/stress incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neck and low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flare up of hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Buttox pain (Nervous system disorders) | 0 (0) | 1 (1) — Buttocks pain; possibly neuritis secondary to BMP
Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator may not submit the results of the study for publication, without the sponsor's prior permission.